CLINICAL TRIAL: NCT04870658
Title: Patient's Perception of Complications in Implantology. Prospective Multicenter Study.
Brief Title: Patient's Perception of Complications in Implantology.
Status: Completed | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: COMPLI
Record Dates: First submitted 2021-04-25; First posted 2021-05-03 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Dental Implant Failed; Dental Prosthesis Failure
Keywords: Complication; Implant dentistry

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complication: Any patients with biological or mechanical complication in dental implant treatment.
  Interventions: Procedure: Dental implant treatment

INTERVENTIONS:
Procedure: Dental implant treatment — Patients who receive one o more dental implant treatment to restore oral function.
  Other Names: Dental implant prosthesis

SUMMARY:
To assess the influence that the complications of implant treatment have on the patient's perception and satisfaction on treatment.

DETAILED DESCRIPTION:
The study is carried out in 5 dental centers with similar socio-professional characteristics.

The perception of patients with complications in implantology will be evaluated using a questionnaire.

All patients who present some type of complication in a dental treatment with implants will be included. Patients will be included both if they are aware of the complication, that is, they come to the consultation for it, and patients who are diagnosed with a complication in a routine check-up.

Patients will be informed of the complication and before explaining the treatment possibilities, their inclusion in the study will be formalized by signing the Informed Consent document.

Subsequently, they must fill out a questionnaire consisting of 5 questions about their perception of the complication and its influence on their quality of life.

The researcher will record the technical data of the implant treatment as well as the patient's responses in the Data Table.

After collecting a sufficient number of data, around 400 patients, the collaborating researchers will send their corresponding data tables to the main researcher who will be in charge of the statistical analysis together with obtaining the results.

ELIGIBILITY:
Inclusion Criteria:

Patients form 18 to 95 years old. Patients with dental implants supporting one o more implant prosthesis. Patients presenting one treatment complication affecting either dental implant or implant prothesis.

Exclusion Criteria:

Patients who does not accept informed consent and do not want to fill the questionnaire.

Patients with cognitive impairment. Patients under psychiatric treatment.

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female.
Study Population: All the patients who present dental implant complication in any of the center in the study.
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Patient´s pain perception | Day 0
  The degree of pain perceived by the patient after the onset of the complication by Numeric Rating Scale (NRS) form 0 to 10, being 0 "No pain" and 10 "Very painful".
Functional impairment | Day 0
  The impact of complication on functional impairment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "Not affected" and 10 "Very affected".
Degree of Concern | Day 0
  The degree of concern that the complication generates in the patient by Numeric Rating Scale (NRS) form 0 to 10, being 0 "Not concerned" and 10 "Very concerned".
Quality of life (QoL) | Day 0
  Patient perception of the impact of the complication on their quality of life by Numeric Rating Scale (NRS) form 0 to 10, being 0 "Not affected" and 10 "Very affected".
Degree of Confidence | Day 0
  The impact that the complication has had on the patient's confidence in dental implant treatment using a numerical rating scale (NRS) from 0 to 10, with 0 being "Confident that they will not receive any further dental implant treatment" and 10 being "Confident that they will".

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, DDS, Principal Investigator — Aula Dental Avanzada
Locations (1):
- Clínica Dental Esteve, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunello G, Gervasi M, Ricci S, Tomasi C, Bressan E. Patients' perceptions of implant therapy and maintenance: A questionnaire-based survey. Clin Oral Implants Res. 2020 Oct;31(10):917-927. doi: 10.1111/clr.13634. Epub 2020 Jul 26. PMID 32645229
- [Background] Derks J, Hakansson J, Wennstrom JL, Klinge B, Berglundh T. Patient-reported outcomes of dental implant therapy in a large randomly selected sample. Clin Oral Implants Res. 2015 May;26(5):586-91. doi: 10.1111/clr.12464. Epub 2014 Aug 14. PMID 25123298
- [Background] Insua A, Monje A, Wang HL, Inglehart M. Patient-Centered Perspectives and Understanding of Peri-Implantitis. J Periodontol. 2017 Nov;88(11):1153-1162. doi: 10.1902/jop.2017.160796. Epub 2017 May 26. PMID 28548884
- [Background] Karlsson K, Derks J, Wennstrom JL, Petzold M, Berglundh T. Occurrence and clustering of complications in implant dentistry. Clin Oral Implants Res. 2020 Oct;31(10):1002-1009. doi: 10.1111/clr.13647. Epub 2020 Sep 4. PMID 32794289